CLINICAL TRIAL: NCT07255274
Title: Treatment of Overweight and Obesity in Adolescents - Impact of a Sleep Behavioral Intervention - SLEEP-OB
Brief Title: Overweight and Obesity in Adolescents - Sleep Behavioral Intervention
Acronym: SLEEP-OB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Beira Interior (Other)
Responsible Party: Principal Investigator, ana sofia rodrigues ferreira, PhD student, University of Beira Interior
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TID 101794088
Record Dates: First submitted 2025-06-14; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Obesity and Overweight; Sleep Disorder
Keywords: Obesity; Sleep; Behavioral intervention; Adolescents
MeSH Terms: conditions — Obesity; Overweight; Sleep Wake Disorders | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: Open-Label Randomized Clinical Study with a Behavioral Intervention
Who Masked: Outcomes Assessor
Masking Description: Randomization is performed by a researcher not involved in data management.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Standard interventions focused on nutrition, physical activity/sedentary behavior, and other lifestyle aspects.
  Interventions: Other: Standard Obesity Treatment
- Intervention group (Experimental): Standard intervention plus sleep-focused intervention. The sleep intervention will be conducted by psychologists. These monthly sessions, delivered in person or via video call, will be scheduled on the same day as the medical consultation whenever possible. The session planning and objectives are outlined in the study protocol.
  Interventions: Behavioral: Sleep Behavioral Intervention; Other: Standard Obesity Treatment

INTERVENTIONS:
Behavioral: Sleep Behavioral Intervention — Our research team, composed by pediatricians with experience in Obesity and Adolescent Medicine, and clinical psychologists with experience in Sleep, Obesity, and Cognitive Behavioral Therapy (CBT), developed a specific manual for this project: "Behavioral Sleep Intervention - SLEEP-OB - Therapist Support Manual." The manual was adapted based on CBT models for adults and adolescents with insomnia and on CBT for adolescents with other sleep disorders and comorbidities, namely obesity. The behavioral intervention aims to promote sustainable changes in sleep. It includes behavioral strategies (such as sleep restriction, stimulus control), cognitive strategies (cognitive reappraisal/restructuring, cognitive control, paradoxical intention), mixed strategies (sleep education/hygiene, relaxation), self-monitoring, and problem identification and resolution.
  The intervention will take place over six months, with a total of seven sessions (in-person and by video call).
  Other Names: Sleep intervention; Cognitive Behavioral Therapy for sleep disorders
  Arms: Intervention group
Other: Standard Obesity Treatment — Standard obesity treatment for pediatric obesity according to international guidelines. It comprises pediatric appointments, and usually also nutrition and nursing appointments, every 2 to 3 months. These appointments include an anthropometric evaluation, physical examination and personalized multicomponent behavioral intervention with focus on nutrition, physical activity/sedentary behavior and other lifestyle recommendations. This standard intervention is common for both groups/arms.
  Other Names: treatment as usual

SUMMARY:
Sleep plays a crucial role in energy balance, alongside diet and physical activity. Research has linked poor sleep quality and short sleep duration to obesity and cardiometabolic risk, such as insulin resistance and hypertension. The nature of this association is complex, and several mechanims have been suggested.

Scientific evidence suggests that sleep interventions may provide additional benefits in optimizing the effectiveness of overweight/obesity treatment in pediatric populations. Although some studies have explored this hypothesis, methodological heterogeneity hampers clear interpretation of the results.

The main goal of this clinical trial is is to evaluate the efficacy of a sleep behavioral intervention, combined with standard obesity treatment, in reducing adiposity (measured by BMI z-score, fat mass percentage, or fat-free mass index) in adolescents with overweight or obesity.

This randomized controlled trial will compare a control group receiving treatment as usual (or standard obesity treatment) with an intervention group receiving treatment as usual plus a sleep behavioral intervention.

Participants will be randomized into two groups: intervention and control. Throughout the study period, all medical consultations will include standard interventions focused on nutrition, physical activity/sedentary behavior, and other lifestyle factors. The sleep-focused intervention will be delivered by psychologists.

Participants will attend clinic visits every two months during the 6-month intervention period, and every three months during the subsequent 6-month follow-up period.

DETAILED DESCRIPTION:
A randomized controlled trial (open-label, behavioral intervention) will be conducted at ULS Cova da Beira and Hospital CUF Porto, enrolling 126 adolescents (ages 13-17) diagnosed with overweight or obesity and poor sleep quality. Participants will be randomized into two groups: the intervention group (sleep behavioral intervention plus treatment as usual) and the control group (treatment as usual).

In addition to the primary aim, the researchers will evaluate several secondary outcomes, including the efficacy of the intervention in relation to: cardiometabolic risk, sleep patterns, eating patterns, physical activity level, emotional well-being/self-compassion, quality of life, leptin and ghrelin levels, and tryptophan and melatonin metabolism.

Throughout the study period, all medical consultations will include standard multicomponent behavioral intervention. The sleep behavioral intervention will be conducted by psychologists.

The intervention consists of seven cognitive-behavioral therapy (CBT) sessions over six months, focusing on sleep hygiene, self-monitoring, stimulus control, cognitive therapy, and relaxation techniques.

Data collection and analysis will include objective sleep assessment using actigraphy and a level 3 ambulatory sleep study. Blood samples will be collected at baseline, six months, and twelve months to analyze metabolic markers. From the samples collected at months 0 and 6, a portion will be appropriately stored for additional analysis at an external facility to quantify leptin, ghrelin, and tryptophan pathway metabolites.

Anthropometric and clinical assessments will include measurements of body mass index (BMI), waist circumference, body composition, and blood pressure. Validated questionnaires will be used to evaluate sleep patterns, eating behaviors, physical activity, quality of life, emotional well-being, and self-compassion.

It is anticipated that the sleep behavioral intervention combined with standard treatment will be more effective than standard treatment alone not only in reducing adiposity, but also in improving cardiometabolic risk, sleep patterns, eating patterns, physical activity, emotional well-being, self-compassion, and in regulating hormonal and metabolic pathways including ghrelin, leptin, and the tryptophan-melatonin axis, as outlined in the study hypotheses

The study also aims to clarify the role of ghrelin and leptin levels, as well as the tryptophan pathway, in the interaction between sleep and obesity and in the effects of the intervention

Emotional well-being and self-compassion are expected to mediate the response to obesity intervention and the sleep-obesity relationship, potentially influencing or influenced by the tryptophan metabolic pathway, particularly serotonin levels.

By deepening the knowledge about the relationship between sleep and obesity, this research may contribute to optimize interventions for pediatric obesity, which would have an unequivocal positive impact.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent from legal guardians and assent/consent from the adolescent;
2. Age between 13 and 17 years at the time of consent;
3. Diagnosis of overweight (BMI z-score > 1 and ≤ 2) or obesity (BMI z-score > 2), according to WHO criteria;
4. Sleep deprivation or poor sleep quality, based on the initial screening questionnaire.

Exclusion Criteria:

1. Secondary obesity (e.g., hypothalamic, genetic, or endocrine causes);
2. Comorbid psychiatric or neurological disorders (e.g., epilepsy, autism spectrum disorder) that affect sleep;
3. Current treatment with selective serotonin reuptake inhibitors (SSRIs) or other medications affecting sleep.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Estimated)
Dates: Start 2025-06-03 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
BMI z-score at 6 months | 6 months
  Variation between Visit 1 (baseline) and Visit 4 (end of the intervention). Weight (in kilograms) and height (in meters) will be used to calculate BMI in kg/m2. Then, BMI z-score will be calculated by WHO Anthroplus software 3.2.2.
BMI at 6 months | 6 months
  Variation between Visit 1 (baseline) and Visit 4 (end of the intervention). Weight (in kilograms) and height (in meters) will be used to calculate BMI in kg/m2.
Fat mass percentage at 6 months | 6 months
  Variation between Visit 1 (baseline) and Visit 4 (end of the intervention). Fat mass percentage (%FM) assessed using bioelectrical impedance analysis with InBody 270®.
Fat-free mass index at 6 months | 6 months
  Variation between Visit 1 (baseline) and Visit 4 (end of the intervention). FFMI (kg/ m2) calculated using FFM (in kilograms) and height (in meters).

SECONDARY OUTCOMES:
Participants achieving a BMI reduction ≥5% | 6 months and 12 months
  Percentage of participants achieving a BMI reduction ≥5% between Visit 1 and Visit 4, and between Visit 1 and Visit 6.
Participants achieving a BMI reduction ≥10% | 6 months and 12 months
  Percentage of participants achieving a BMI reduction ≥10% between Visit 1 and Visit 4, and between Visit 1 and Visit 6.
Change in Waist circumference centile | 6 months and 12 months
  Variation between Visit 1 and Visit 4, and between Visit 1 and Visit 6. waist circumference in centimeters, and centiles according to Sharma AK, et al. Pediatr Res. 2015.
Fat mass percentage at 12 months | 12 months
  Variation between Visit 1 (baseline) and Visit 6 (end of the follow-up). Fat mass percentage (%FM) assessed using bioelectrical impedance analysis with InBody 270®.
Fat-free mass index at 12 months | 12 months
  Variation between Visit 1 (baseline) and Visit 6 (end of the follow-up). FFMI (kg/ m2) calculated using FFM (in kilograms) and height (in meters).
BMI z-score at 12 months | 12 months
  Variation between Visit 1 (baseline) and Visit 6 (end of the follow-up). Weight (in kilograms) and height (in meters) will be used to calculate BMI in kg/m2. Then, BMI z-score will be calculated by WHO Anthroplus software 3.2.2.
BMI at 12 months | 12 months
  Variation between Visit 1 (baseline) and Visit 6 (end of the follow-up). Weight (in kilograms) and height (in meters) will be used to calculate BMI in kg/m2.
Change in Waist-to-height Ratio | 6 months and 12 months
  Variation between Visit 1 and Visit 4, and between Visit 1 and Visit 6.
Change in C-reactive protein | 6 months and 12 months
  Variation between Visit 1 and Visit 4, and between Visit 1 and Visit 6.
Change in Fasting Lipid: Total Cholesterol | 6 months and 12 months
  Variation between Visit 1 and Visit 4, and between Visit 1 and Visit 6.
Change in Fasting Lipid: LDL-cholesterol | 6 months and 12 months
  Variation between Visit 1 and Visit 4, and between Visit 1 and Visit 6.
Change in Fasting Lipid: HDL-cholesterol | 6 months and 12 months
  Variation between Visit 1 and Visit 4, and between Visit 1 and Visit 6.
Change in Fasting Lipid: Triglycerides | 6 months and 12 months
  Variation between Visit 1 and Visit 4, and between Visit 1 and Visit 6.
Change in centiles of Systolic and Diastolic Blood Pressure | 6 months and 12 months
  Variation between Visit 1 and Visit 4, and between Visit 1 and Visit 6. Blood pressure measured and centiles according to the American Academy of Pediatrics.
Change in HbA1c | 6 months and 12 months
  Variation between Visit 1 and Visit 4, and between Visit 1 and Visit 6.
Change in Glycaemic Category | 6 months and 12 months
  Variation between Visit 1 and Visit 4, and between Visit 1 and Visit 6. Number of participants in glycaemic categories, "normoglycaemia, pre-diabetes and type 2 diabetes (T2DM)" 2 are presented. These categories were set as per the following criteria: 1) Normoglycaemia: fasting plasma glucose (FPG) <100 mg/dL and/or HbA1c <5.7%. 2) Pre-diabetes: FPG 100-125 mg/dL (both inclusive) or HbA1c 5.7-6.4% (both inclusive). 3) Type 2 diabetes (T2DM): FPG ≥126 mg/dL and/or HbA1c ≥6.5%
Change in HOMA-B | 6 months and 12 months
  Variation between Visit 1 and Visit 4 and between Visit and Visit 6. HOMA-B was calculated as: Beta-cell function (%) = 20·fasting insulin[mU/L]/(FPG[mmol/L]-3.5).
Change in HOMA-IR | 6 months and 12 months
  Variation between Visit 1 and Visit 4 and between Visit and Visit 6. HOMA-IR was calculated as: Insulin resistance (%) = fasting insulin [mU/L] x FPG [mmol/L]/ 22.5. R
Change in Continuous metabolic syndrome score | 6 months and 12 months
  Variation between Visit 1 and Visit 4 and between Visit and Visit 6. Calculation according to Vukovic R, et al. PLoS One. 2017 Dec 6;12(12):e0189232.
Change in Sleep quality | 6 months and 12 months
  Sleep quality assessed by the Pittsburgh Sleep Quality Index, at Visit 1and Visit 4, and at Visit 6.
Change in sleep quality - actigrafy | 6 months
  Sleep quality assessed by actigraphy and sleep diary, at Visit 1and Visit 4.
Change in Respiratory Sleep disorder | 6 months
  Respiratory sleep disorder assessed by the Pediatric sleep questionnaire at Visit 1and Visit 4.
Change in Diet Quality | 6 months
  Mediterranean Diet Quality assessed with KIDMED questionnaire, at Visit 1 and Visit 4.
Change in Eating behavior | 6 months
  MEating behavior assessed with Eating Attitudes Test questionnaire, at Visit 1 and Visit 4.
Change in emotional well-being | 6 months
  At Visit 1 and Visit 4: Emotional well-being assessed through the WHO-5.
Change in Quality of life | 6 months
  At Visit 1 and Visit 4: Quality of life evaluated with the KIDSCREEN 52 questionnaire.
Change in self-compassion | 6 months
  At Visit 1 and Visit 4: Self-compassion evaluated with the Self-Compassion Scale for adolescents.
Change in Physical activity | 6 months
  Physical activity assessed with International Physical Activity Questionnaire for Adolescents, at Visit 1 and Visit 4.
Change in Physical activity - actigraphy | 6 months
  Physical activity assessed by actigraphy, at Visit 1 and Visit 4.

OTHER OUTCOMES:
Tryptophan pathway metabolites measurement | 6 months
  Levels of tryptophan, kynurenine, serotonin, and melatonin in plasma samples, by metabolomic analysis/ liquid chromatography, at baseline (Visit 1) and after the Intervention (Visit 4).
Leptin and ghrelin levels | 6 months
  Levels of leptin and ghrelin will be measured in plasma samples using enzyme-linked immunosorbent assay (ELISA) at baseline (Visit 1) and after the intervention (Visit 4).

CONTACTS AND LOCATIONS:
Locations (2):
- Portugal (2):
  - Unidade Local de Saúde Cova da Beira, Covilha
  - Hospital CUF Porto, Porto

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be shared upon request, provided that all identifying information is removed to safeguard participant anonymity. This process upholds the confidentiality and privacy of participants, fully complying with ethical and legal standards for data protection.
Supporting Information: Study Protocol, SAP
Time Frame: June 2026 to June 2027
Access Criteria: The data supporting the findings of this study will be available upon request from the corresponding author. Each request will be reviewed by the research team and the Ethics Committees that approved the study to ensure compliance with ethical standards.